CLINICAL TRIAL: NCT05221502
Title: A Multicenter, Phase 2b/c, Open-label, Randomized, Dose-finding Trial to Evaluate the Safety and Efficacy of a 4 Month Regimen of OPC-167832 in Combination With Delamanid and Bedaquiline in Subjects With Drug-susceptible Pulmonary Tuberculosis in Comparison With Standard Treatment
Brief Title: Safety and Efficacy Evaluation of 4-month Regimen of OPC-167832, Delamanid and Bedaquiline in Participants With Drug-Susceptible Pulmonary TB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 323-201-00006
Record Dates: First submitted 2021-08-20; First posted 2022-02-03 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary TB
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — OPC-67683; bedaquiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Delamanid + Bedaquiline + OPC-167832 10 mg (Experimental): Participants will receive a combination regimen of delamanid, 300 mg, oral tablets, once daily (QD), bedaquiline, 400 mg, oral tablets, QD for 2 weeks, then 200 mg, thrice weekly (TIW) and OPC-167832, 10 mg, oral tablets, QD for a total of 17 weeks.
  Interventions: Drug: Delamanid + Bedaquiline + OPC-167832 10 mg
- Delamanid + Bedaquiline + OPC-167832 30 mg (Experimental): Participants will receive a combination regimen of delamanid, 300 mg, oral tablets, QD, bedaquiline, 400 mg, oral tablets, QD for 2 weeks, then 200 mg, TIW and OPC-167832, 30 mg, oral tablets, QD for a total of 17 weeks.
  Interventions: Drug: Delamanid + Bedaquiline + OPC-167832 30 mg
- Delamanid + Bedaquiline + OPC-167832 90 mg (Experimental): Participants will receive a combination regimen of delamanid, 300 mg, oral tablets, QD, bedaquiline, 400 mg, oral tablets, QD for 2 weeks, then 200 mg, TIW and OPC-167832, 90 mg, oral tablets, QD for a total of 17 weeks.
  Interventions: Drug: Delamanid + Bedaquiline + OPC-167832 90 mg
- Rifampin, Isoniazid, Ethambutol, and Pyrazinamide (RHEZ) (Active Comparator): Participants will receive RHEZ, orally, QD for 8 weeks followed by 18 weeks of rifampin and isoniazid for a total of 26 weeks.
  Interventions: Drug: RHEZ

INTERVENTIONS:
Drug: Delamanid + Bedaquiline + OPC-167832 10 mg — Delamanid (300 mg QD) + Bedaquiline (400 mg QD x 2 weeks, then 200 mg TIW) + OPC-167832 (10 mg QD) for 17 weeks
  Arms: Delamanid + Bedaquiline + OPC-167832 10 mg
Drug: Delamanid + Bedaquiline + OPC-167832 30 mg — Delamanid (300 mg QD] + Bedaquiline (400 mg QD x 2 weeks, then 200 mg TIW) + OPC-167832 (30 mg QD) for 17 weeks
  Arms: Delamanid + Bedaquiline + OPC-167832 30 mg
Drug: Delamanid + Bedaquiline + OPC-167832 90 mg — Delamanid (300 mg QD) + Bedaquiline (400 mg QD x 2 weeks, then 200 mg TIW) + OPC-167832 (90 mg QD) for 17 weeks
  Arms: Delamanid + Bedaquiline + OPC-167832 90 mg
Drug: RHEZ — RHEZ for 8 weeks followed by 18 weeks of rifampin and isoniazid (for a total of 26 weeks)
  Arms: Rifampin, Isoniazid, Ethambutol, and Pyrazinamide (RHEZ)

SUMMARY:
This trial will assess the safety and efficacy of OPC-167832 combined with delamanid and bedaquiline in participants with drug-susceptible tuberculosis (DS-TB) administered for 17 weeks compared to rifampin, isoniazid, ethambutol, pyrazinamide (RHEZ) administered for 26 weeks.

DETAILED DESCRIPTION:
Eligible participants for this study have a diagnosis of pulmonary DS-TB.

This is a Phase 2b/c multicenter, open-label, randomized, dose-finding study, consisting of up to 26 weeks of treatment period.

Following a screening period of up to 14 days, eligible participants will be randomized in the study.

Randomization will be stratified by presence of bilateral cavitation on screening chest x-ray (yes or no). After the end of the treatment period, participants will be followed until 12 months post randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written, informed consent prior to initiation of any trial-related procedures or treatments, and able, in the opinion of the investigator, to comply with all the requirements of the trial.
2. Male or female participants between 18 and 65 years of age (inclusive) at the screening visit.
3. Body weight ≥ 35.0 kg at the screening visit.
4. Newly diagnosed, rifampin and isoniazid susceptible (on the screening sample) pulmonary TB.
5. Able to spontaneously produce sputum.
6. Females of childbearing potential (FOCBP) must agree to use 2 different approved methods of birth control or remain abstinent throughout their participation in the trial and for 12 weeks after the last dose of IMP or dose of RHEZ.
7. Male participants must agree to use 2 different approved methods of birth control or remain abstinent throughout their participation in the trial and for 12 weeks after the last dose of IMP or RHEZ.

Exclusion Criteria:

1. Participants are known or suspected of having resistance to rifampin, isoniazid, ethambutol, pyrazinamide, DLM, or BDQ either confirmed by the laboratory, or based on epidemiological history, at screening.
2. Evidence of clinically significant metabolic (for example, including ongoing or current hypokalemia [ie, potassium <3.5 mEq/dL at screening]), gastrointestinal, neurological, psychiatric, endocrine or liver (eg, hepatitis B and C) disease; malignancy; or other abnormalities (other than the indication being studied).
3. History of, or current, clinically relevant cardiovascular disorder such as heart failure, coronary heart disease, uncontrolled hypertension, arrhythmia or symptom strongly suggestive of such a problem (for example, syncope or palpitations), tachyarrhythmia or status after myocardial infarction.
4. Known bleeding disorders or family history of bleeding disorders.
5. Any diseases or conditions in which the use of DLM, BDQ, OPC 167832, rifampin, isoniazid, pyrazinamide, or ethambutol is contraindicated.
6. Any prior treatment for M tuberculosis within the past 2 years.
7. Any treatment with a drug active against M tuberculosis (eg, quinolones) within the 3 months prior to screening.
8. Clinical evidence of severe extrapulmonary TB (eg, miliary TB, abdominal TB, urogenital TB, osteoarthritic TB, TB meningitis).
9. Evidence of pulmonary silicosis, lung fibrosis, or other lung condition considered as severe by the investigator (other than TB). In particular, any underlying condition that could interfere with the assessment of x-ray images, sputum collection, or interpretation of sputum findings, or otherwise compromise the subject's participation in the trial.
10. Any renal impairment characterized by creatinine clearance/estimated glomerular filtration rate (eGFR) of < 60 mL/min/1.73 m2, or hepatic impairment characterized by alanine transaminase or aspartate transaminase > 2.0 × upper limit of normal of the clinical laboratory reference range or bilirubin > 2.0 × upper limit of normal of the clinical laboratory reference range, at screening.
11. Screening glucose (nonfasting) ≥ 200 mg/dL or glycosylated hemoglobin (HbA1c) ≥ 6.5%.
12. QTcF > 450 msec in male participants (> 470 msec in female participants), atrioventricular block II or III, bi-fasicular block, at screening or current or history of clinically significant ventricular arrhythmias. Other ECG abnormalities, if considered clinically significant by the investigator.
13. Participants receiving any of the prohibited medications (see Section 6.5.1) within the specified periods or who would be likely to require prohibited concomitant therapy during the trial.
14. Female participants who are breast-feeding or who have a positive pregnancy test result prior to receiving the first dose of IMP or RHEZ on Day 1.
15. Current history of significant drug and/or alcohol abuse that is likely to result in poor adherence to trial requirements or that would pose a risk to the participant's well-being during the course of the trial.
16. History of current hepatitis or carriers of hepatitis B surface antigen (HBsAg) and/or anti hepatitis C virus (HCV).
17. Participants who test positive for cocaine or other drugs of abuse (excluding known prescription stimulants and other prescribed medications and marijuana) at screening are excluded. Detectable levels of alcohol, marijuana, barbiturates, or opiates in the drug screen are not exclusionary if, in the investigator's documented opinion, the participant does not meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition criteria for moderate to severe substance use disorder and the positive test does not signal a clinical condition that would impact the safety of the participant or interpretation of the trial results, and participation is agreed to by the medical monitor prior to treatment.
18. History of having taken an investigational drug within 30 days preceding trial entry.
19. A history of difficulty in donating blood.
20. Donation of blood or plasma within 30 days prior to dosing.
21. History of serious mental disorders that, in the opinion of the investigator, would exclude the participant from participating in this trial.
22. Any known prior exposure to OPC-167832, DLM, or BDQ.
23. Participants with significant medical comorbidities that in the opinion of the investigator, should not participate in the trial.
24. Participants with Karnofsky score < 60 will be excluded from the trial.
25. Participants testing positive for active severe acute respiratory syndrome coronavirus (SARS-CoV-2) infection at screening.
26. Participants with HIV co infection not on a stable anti-retroviral regimen consisting of tenofovir, emtricitabine/ lamivudine, dolutegravir (ie > 3 months), or who have a detectable viral load, or who have a CD4 count < 350 cells/mm3 will be excluded from the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-05-19 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events | Baseline to 12 months post randomization
  Incidence of TEAEs: all TEAEs, TEAEs by severity, TEAEs potentially causally related to the IMP or trial medication, TEAEs with an outcome of death or trial medication, Serious TEAEs, TEAEs leading to discontinuation of the IMP or trial medication
Incidence of potentially clinically significant changes of laboratory tests from baseline and abnormalities in the vital signs, physical examinations, electrocardiograms (ECGs) at each visit were assessed and at end of study. | Baseline to 12 months post randomization
  Incidence of potentially clinically significant changes from baseline and abnormalities in the parameters below, at each visit were assessed and at end of study:
  Lab Tests: Hematology, Clinical Chemistry, CD4 Count, Urinalysis Vital Signs: systolic and diastolic blood pressure (mmHg), heart rate (beats/min), respiratory rate (breaths/min), body temperature (C), weight (kg) and body mass index (kg/m2)
  Physical exam include examination of the abdomen; extremities; head, eyes, ears, nose (HEENT); neurological; skin and mucosae; thorax; urogenital; audiometry assessment and visual assessment.
  ECGs:
  ECG PR interval (msec) ECG QTc interval (msec) ECG arrhythmia
Number of participants with a grade 3 or higher AE | Baseline to 12 months post randomization
  The proportion of subjects with a grade 3 or higher AE
Number of all cause Treatment Discontinuation | Baseline to 12 months post randomization
  Rate of All Cause Treatment Discontinuation
Sputum culture conversion (SCC) in Mycobacteria Growth Indicator Tube® (MGIT) | Baseline to End of Treatment Period - Week 17 and Week 26
  The proportion of subjects achieving sputum culture conversion (SCC) in Mycobacteria Growth Indicator Tube® (MGIT) (Sputum culture conversion occurs when a subject has the first of 2 visits of at least 1 week apart (±4 days) with sputum cultures negative and without a positive sputum culture result in between).

SECONDARY OUTCOMES:
Proportion of participants who achieve SCC in MGIT by 8 weeks of treatment | Baseline to Week 8
  Proportion of subjects who achieve SCC.
Time to detection of MGIT cultures | Baseline to 12 months post randomization
  Change in time to detection, in days, of MGIT liquid culture results
Proportion of participants who convert sputum LAM to negative by 8 weeks of treatment and by end of treatment | End of Treatment Period - Week 17 and Week 26
  The proportion of subjects who convert sputum LAM concentrations from positive to negative by 8 weeks of treatment and by end of treatment
Proportion of participants who develop drug resistance | Baseline to 12 months post randomization
  Proportion of subjects whose sputum cultures test "resistant" to any drugs in the treatment regimens during the treatment period.
Time to Sputum Culture Conversion (SCC) of each treatment group. | Baseline to 12 months post randomization
  To compare time to SCC, in days, of each treatment group.

OTHER OUTCOMES:
Assess the positron emission tomography/computerized axial tomography (PET/CT) imaging response over the course of treatment | Baseline to Week 26
  Positron emission tomography/computerized axial tomography (PET/CT) imaging changes over the course of treatment, using quantitative scan assessment.
Evaluate the ribosomal ribonucleic acid synthesis ratio (RS ratio) decline in sputum | Baseline to 12 months post randomization
  The decline of ribosomal ribonucleic acid synthesis ratio (RS ratio - a ratio of spacers between the mRNA) in sputum over the course of trial.
Assess whole blood transcriptomic signatures previously associated with TB cure from serum | Screening to 12 months post randomization
  The change in whole blood transcriptomic signatures over the course of treatment will be evaluated using ROC curves for association with microbiological and clinical response.
The proportion of participants with favorable outcome at 12 months post randomization | Baseline to 12 months post randomization
  The proportion of subjects with favorable outcome as compared to the 6 months post end of treatment and at 12 months post randomization.
Number of participants with relapse at 12 months post randomization | Baseline to 12 months post randomization
  Proportion of participants with relapse at 12 months post randomization.

CONTACTS AND LOCATIONS:
Locations (6):
- South Africa (6):
  - Aurum Institute - Tembisa Clinical Research Centre, Tembisa, Gauteng
  - TASK Applied Science, Brooklyn Chest Hospital Premises, Cape Town
  - University of CapeTown Lung Center Institute, Cape Town
  - Themba Lethu Clinic Clinical HIV Research Unit (CHRU), Johannesburg
  - Perinatal HIV Research Unit Tshepong Hospital Complex, Klerksdorp
  - Setshaba Research Center, Pretoria

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

REFERENCES:
- [Derived] Dawson R, Diacon AH, Takuva S, Liu Y, Zheng B, Karwe V, Hafkin J. Quabodepistat in combination with delamanid and bedaquiline in participants with drug-susceptible pulmonary tuberculosis: protocol for a multicenter, phase 2b/c, open-label, randomized, dose-finding trial to evaluate safety and efficacy. Trials. 2024 Jan 19;25(1):70. doi: 10.1186/s13063-024-07912-5. PMID 38243296